CLINICAL TRIAL: NCT06692400
Title: The Impact of Endotracheal Suctioning on Pain, Hypoxia, and Oxidative Stress Biomarkers in Intubated Adult ICU Patients: A Controlled Trial
Brief Title: The Effects of Endotracheal Suctioning on Pain and Serum Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5240556
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Intensive Care Unit ICU; Intubation; Critical Illness; Mechanical Ventilation; Pain Measurement; Pain, Procedural; Oxidative Stress; Hypoxia; Biomarkers / Blood; Adult; Uric Acid; Sepsis; COVID; Influenza; Pneumonia
MeSH Terms: conditions — Critical Illness; Pain, Procedural; Hypoxia; Sepsis; Influenza, Human; Pneumonia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The lab technician who results the labs will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants who undergo endotracheal tube (ETT) suctioning. (Experimental): Participants will receive ETT suctioning as part of routine care.
  Interventions: Procedure: endotracheal tube suctioning
- Participants who do not undergo ETT suctioning during the observation period. (No Intervention): Participants will not receive ETT suctioning during the observation periood.

INTERVENTIONS:
Procedure: endotracheal tube suctioning — Endotracheal tube suctioning occurs as part of normal care for intubated patients. This procedure will serve as the painful procedure to assess CPOT and biomarkers of hypoxia and oxidative stress.
  Arms: Participants who undergo endotracheal tube (ETT) suctioning.

SUMMARY:
The goal of this experimental study is to understand if endotracheal tube (ETT) suctioning increases pain and causes stress on the body in intubated adult ICU patients. These patients are already on ventilators, which means they need suctioning to keep their airways clear, but this procedure may be uncomfortable and cause stress.

The main questions this study aims to answer are:

Does ETT suctioning raise pain levels as measured by the Critical-Care Pain Observation Tool (CPOT)? Does ETT suctioning increase certain chemicals in the blood (hypoxanthine, xanthine, and uric acid) that show stress and lack of oxygen in the body? Researchers will compare patients who have ETT suctioning (intervention group) with those who do not have suctioning during the study period (control group) to see if there are differences in pain and blood markers of stress.

Participants will:

Have pain measured before and after suctioning using the CPOT. Have blood samples taken from an existing line at three time points: 5 minutes before, 5 minutes after, and 30 minutes after suctioning.

Provide demographic information (like age, gender, and diagnosis) from medical records.

This research will help improve how pain is managed for ICU patients who cannot speak for themselves, potentially leading to better pain relief methods in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years and older)
* Current diagnosis of flu, pneumonia, COVID, or sepsis
* Intubated and receiving mechanical ventilation.
* Have arterial lines placed
* Require endotracheal suctioning as part of their care

Exclusion Criteria:

* Patients receiving neuromuscular blocking agents
* Contraindications for blood draws (hemoglobin levels below 8.0 g/dL; Jehovah's Witness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Impact of ETT suctioning on subject pain level | Change between baseline CPOT score and 30-minutes post suctioning CPOT score.
  The Critical-Care Pain Observation Tool (CPOT) is a composite measurement used to assess pain in non-verbal ICU patients by evaluating four behavioral indicators: facial expression, body movements, muscle tension, and ventilator compliance (for intubated patients) or vocalization (for non-intubated patients). Each indicator is scored from 0 (no pain behavior) to 2 (intense pain behavior), resulting in a total score from 0 to 8. Higher scores indicate higher pain levels, guiding clinicians in pain management. For example, a score of 0 indicates no pain, while a score of 2 in any category suggests more severe pain, prompting possible adjustments in analgesic care.
Impact of ETT suctioning on subject serum markers of hypoxia and oxidative stress (Hypoxanthine). | Change between baseline serum marker blood draw and 30-minutes post suctioning serum marker blood draw
  Serum markers will be obtained via arterial line blood draw 5 minutes pre-ETT suctioning and again post-ETT suctioning. Normal blood concentrations of hypoxanthine in healthy adult individuals are less than 5 µmol. Levels greater than 5 µmol indicate hypoxia and oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Johnston Taylor, PhD, FAAN, Principal Investigator — Loma Linda University School of Nursing
Locations (1):
- Loma Linda University Medical Center Troesh Medical Campus, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Following the completion of this experiment, specific IPD will be shared in de-identified form to support transparency, replication, and further research:
  Demographic data (age, gender, diagnosis) relevant to understanding participant characteristics.
  Pain assessment scores (Critical-Care Pain Observation Tool [CPOT] scores) collected at baseline, 5 minutes, and 30 minutes post-suctioning.
  Biochemical marker levels for hypoxanthine, xanthine, and uric acid, measured at the same time points.
  The IPD will be accessible to qualified researchers upon reasonable request and after ethical and institutional review, following institutional and regulatory guidelines for data sharing. Data will be shared primarily for the purposes of publication in peer-reviewed journals and to facilitate future studies that may enhance supportive care protocols for ICU patients. The data will be available through an encrypted institutional repository to ensure participant confidentiality and data security.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 6 months after publication with no end date
Access Criteria: Who: Researchers with a verified institutional affiliation and approval from their IRB or ethics committee, as applicable. Requests from researchers affiliated with reputable institutions will be reviewed by the primary investigator and the Loma Linda University Health IRB.
  What: De-identified IPD, including Demographic data (age, gender, diagnosis); CPOT pain scores recorded at baseline, 5 minutes, and 30 minutes post-suctioning; Biochemical marker levels (hypoxanthine, xanthine, uric acid) measured at the same time points.
  Relevant study protocols and descriptions of data collection and processing procedures.
  How: Interested researchers must submit a data access request, including a brief research proposal, institutional affiliation, and IRB or ethics approval. Approved researchers will sign a Data Use Agreement (DUA) outlining the terms of use, data confidentiality requirements, and publication guidelines. Access will be provided through a secure, encrypted institutional repository.

REFERENCES:
- [Background] Angeles DM, Boskovic DS, Tan JC, Shih W, Hoch E, Forde D, Phillips RM, Hopper A, Deming DD, Goldstein M, Truong G, Febre A, Pegis P, Lavery A, Kadri M, Banerji A, Mousselli I, Farha V, Fayard E. Oral dextrose reduced procedural pain without altering cellular ATP metabolism in preterm neonates: a prospective randomized trial. J Perinatol. 2020 Jun;40(6):888-895. doi: 10.1038/s41372-020-0634-0. Epub 2020 Feb 26. PMID 32103160